CLINICAL TRIAL: NCT05660421
Title: A Phase II Study of Itacitinib in Patients With Steroid Refractory Immune Related Adverse Events Arising From Immune Checkpoint Inhibitors
Brief Title: Itacitinib for the Treatment Steroid Refractory Immune Related Adverse Events Arising From Immune Checkpoint Inhibitors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual and funding
Sponsor: Douglas Johnson (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor-Investigator, Douglas Johnson, Associate Professor of Medicine, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICCCTT2193; NCI-2022-09649 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2022-11-30; First posted 2022-12-21 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — itacitinib; Adrenal Cortex Hormones; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (itacitinib) (Experimental): Patients receive itacitinib PO and corticosteroids PO or IV. Patients may undergo endoscopy and skin biopsy throughout the study. Patients also undergo blood collection throughout the study.
  Interventions: Drug: Itacitinib; Drug: Corticosteroid; Procedure: Endoscopic Procedure; Procedure: Skin biopsy; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Itacitinib — Given by mouth
Drug: Corticosteroid — Given by mouth or by vein
Procedure: Endoscopic Procedure — Undergo endoscopic procedure
Procedure: Skin biopsy — Undergo skin biopsy
Procedure: Biospecimen Collection — Undergo collection of blood and stool

SUMMARY:
This phase II trial tests how well itacitinib works in in patients with immune related adverse events (irAEs) arising from immune checkpoint inhibitors (ICI) that do not respond to steroids (steroid refractory). Steroids are the usual treatment for these side effects. However, sometimes steroids do not improve or fix the side effects. Giving itacitinib may be effective in treating patients with known or suspected problems coming from ICIs, that do not resolve or improve with steroids, by reducing the patients immune system response that can cause the irAEs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To define the rate of improvement of steroid-refractory immune related adverse events (irAEs) in patients treated with ICI at 28 days.

SECONDARY OBJECTIVES:

I. To define whether anti-tumor activity is preserved (response rate, progression free survival [PFS], T cell populations and function in the tumor).

II. To assess freedom from hospitalization and any grade improvement at 14 and 28 days.

III. To assess rate of therapy escalation (increased dose of steroids, other immunosuppressant) by day 60 follow up.

IV. To define cancer-specific and toxicity-specific survival at 6 months. V. To define the rate of improvement of steroid-refractory irAEs in patients treated with ICI at any time, and at 60 days (defined as improvement to Common Terminology Criteria for Adverse Events [CTCAE] Grade 0-1).

VI. To define the proportion of patients able to be tapered off steroids at Day 29 and at Day 30 follow up.

VII. To define the safety of itacitinib in patients with steroid-refractory irAEs.

OUTLINE:

Patients receive itacitinib orally (PO) and corticosteroids PO or intravenously (IV) on study. Patients may undergo endoscopy and skin biopsy throughout the study. Patients also undergo blood collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal participant care.
* Must be willing and able to comply with scheduled visits, treatment schedule,laboratory tests, biopsies, and other requirements of the study.
* Must have received at least one immune checkpoint inhibitor (ICI) therapy either as single agent(s) or in combination(s), including but not limited to nivolumab, ipilimumab, pembrolizumab, cemiplimab, atezolizumab, durvalumab, or avelumab.
* Must experience at least one Grade 2, 3 or 4 (CTCAE Version 5.0) toxicity/immune-related adverse event (irAE) attributed to immune checkpoint inhibitor (ICI) therapy as diagnosed by the patient's study physician. This may be established by clinical, histological, or imaging criteria as defined below:

  * Symptoms must be attributed to an immune-related adverse event (irAE), with no infectious or alternative cause suspected by the patient's study physician.
  * Must be actively experiencing Grade 2+ irAE (at the time of screening) as broadly defined below:

    * Cutaneous toxicity (including skin rash)
    * Colitis/enteritis (As defined by Grade 2+ diarrhea or Grade 2+ colitis (either or both conditions)
  * Pneumonitis
  * Arthritis
  * Hepatitis (As defined by Grade 2+ elevation in AST or ALT (either or both values elevated)
  * Nephritis (As defined by either Grade 2+ elevation in creatinine and/or proteinuria of at least 2+ on urinalysis attributed to ICI)
  * Myocarditis (Given the vague nature of symptomatic myocarditis grading, troponin levels will be primarily used to grade myocarditis,( Troponin >2ng/ml), (Presumed diagnosis of myocarditis (myocardial infarction ruled out clinically)
  * Myositis (Defined as grade 2 myositis symptoms per CTCAE OR grade 2 elevations in creatinine kinase levels)
  * Neurologic toxicity

    * Encephalitis

      * Neurologic symptoms consistent with encephalitis
      * Lumbar puncture and infectious disease consult to rule out infectious etiologies if clinical suspicion for infectious causes
    * Guillain Barre

      * MRI performed to rule out spinal cord compression
      * Neurology consult to confirm diagnosis (or extremely high suspicion)
    * Myasthenia Gravis

      * MRI performed to rule out spinal cord compression and brain metastases
      * Neurology consult to confirm diagnosis (or extremely high suspicion)
  * Pericarditis
  * Vasculitis
  * Gastritis
  * Other toxicities

    * Other steroid refractory toxicities not listed in the above list
    * NOTE: Endocrine toxicities (including hypophysitis, hypopituitarism, hypothyroidism, thyrotoxicosis, immune checkpoint inhibitor-induced diabetes, and primary adrenal insufficiency) will NOT qualify for inclusion.
* Must have received oral or intravenous corticosteroids of at least 50mg per day prednisone equivalent dosing (approximately 1mg/kg daily) for ≥ 48 hours of therapy with worsening or lack of improvement to Grade 2.
* May have been treated with additional immunomodulators (one or more) prior to study entry (e.g. infliximab, mycophenolate mofetil, intravenous immunoglobulin), provided such immunomodulators are discontinued prior to first dose of study therapy.
* Adequate organ and marrow function as defined below:

  * White blood cell (WBC) ≥ 2.0 ×109/L.
  * Neutrophil (ANC) ≥ 1.5 ×109/L.
  * Platelet (PLT) ≥ 75 ×109/L.
  * Hemoglobin (Hgb) ≥ 8.0 g/dL.
  * AST and ALT ≤ 3 x ULN in subjects without hepatic metastases; AST and ALT ≤ 5 x ULN in subjects with hepatic metastases, if AST/ALTelevation is NOT due to ICI-induced hepatitis; (Exception (without or with hepatic metastases): no limit for patients with ICI-induced hepatitis).
  * Total bilirubin ≤ 2 x ULN not due to ICI-hepatitis (except subjects with Gilbert syndrome, where total bilirubin must be < 3.0 mg/dL), (Exception: no limit for patients with ICI-induced hepatitis).
* Reproductive status:

  * Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to the start of study treatment.
  * Women must not be breastfeeding.
  * Women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of study drug treatment and 60 days after the last dose of study treatment or longer if required based on prior immunotherapy received (for example, at least 4-5 months for nivolumab and pembrolizumab).
  * Males who are sexually active with Women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of study treatment and 60 days after the last dose of study drug or longer if required based on prior immunotherapy received.
  * Azoospermic males are exempt from contraceptive requirements. WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements but still must undergo pregnancy testing as described in this section.
  * Investigators shall counsel Women of childbearing potential, and male participants who are sexually active with Women of childbearing potential on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise on the use of highly effective methods of contraception which have a failure rate of < 1% when used consistently and correctly. Women of childbearing potential and men must agree to use adequate contraception (for example, hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of protocol treatment.

Exclusion Criteria:

* Toxicity deemed by patient's study physician to be primarily caused by another etiology (bacterial infection, other anticancer agents, etc.).
* Ongoing serious infection requiring IV antibiotics.
* Prior treatment with a JAK inhibitor within the past 8 weeks before first dose of protocol indicated treatment.
* Known HIV infection with CD4 count < 200. (Testing not required by this study.)
* History or current diagnosis of cardiac disease indicating significant risk of safety for participation in the study, such as uncontrolled or significant cardiac disease, including any of the following:

  * Recent myocardial infarction (within 6 months before first dose of protocol indicated treatment).
  * New York Heart Association Class III or IV congestive heart failure.
  * Unstable angina (within last 6 months before first dose of protocol-indicated treatment).
  * Clinically significant (symptomatic) cardiac arrhythmias per judgment of patient's study physician (e.g., sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker).
  * Uncontrolled hypertension defined as blood pressure persistently above 160 systolic or 100 diastolic despite antihypertensive therapy.
* Known allergies, hypersensitivity, or intolerance to any study medications or excipients.
* History of solid organ transplant or allogeneic stem cell transplant with active graft versus host disease.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug/treatment and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of immune related adverse events (irAE) | Baseline up to 60 days post last dose of itacitinib

SECONDARY OUTCOMES:
Objective response rate | Baseline up to 60 days post last dose of itacitinib
  Will be measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as best response reported by the investigator at scans subsequent to itacitinib therapy and will be obtained descriptively by chart review.
Progression-free survival | Baseline up to 60 days post last dose of itacitinib
  Will be obtained using RECIST 1.1 and obtained descriptively by chart review.
Hospitalization presence | Days 14 and 28
  Need for hospitalization will be recorded.
Need for therapy escalation and presence of steroids | From start of itacitinib to 60 days after stopping itacitinib
  The presence of additional immunosuppression added after starting itacitinib or escalation of steroid dose will be recorded.
Need for therapy escalation and absence of steroids | From start of itacitinib to 60 days after stopping itacitinib
  The absence of additional immunosuppression added after starting itacitinib or escalation of steroid dose will be recorded.
The rate of delayed relapses will be followed. | Baseline up to 60 days post last dose of itacitinib
  Rate of irAEs
The rate of improvement at earlier timepoints will be followed. | Baseline up to 60 days post last dose of itacitinib
  Rate of irAEs
Rate of irAEs | Baseline up to 60 days post last dose of itacitinib
  The rate of ability to resume ICI (in select patients, per study investigator decision) will be followed.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Johnson, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT05660421/ICF_000.pdf